CLINICAL TRIAL: NCT06831500
Title: A Monocentric, Randomized, Double-blind Study to Assess the Feasibility of Conducting a Full-scale Randomized Controlled Trial (RCT) Assessing the Effect of Carbidopa/Levodopa Ratio on Orthostatic Hypotension (OH) in Multiple System Atrophy - Parkinsonian Type (MSA-P) and Parkinson Disease (PD) Patients (CARBIDOH)
Brief Title: Feasibility Study Assessing the Effect of Carbidopa/Levodopa Ratio on Orthostatic Hypotension in Multiple System Atrophy - Parkinsonian Type and Parkinson Disease.
Acronym: CARBIDOH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Julien Bally (Other)
Responsible Party: Sponsor-Investigator, Julien Bally, Principal Investigator and Head of the Movement Disorder Unit in the department of Clinical Neurosciences (CHUV), University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-02568
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-07

CONDITIONS: Multi-system Atrophy - Parkinsonian Type; Orthostatic Hypotension, Dysautonomic; Parkinson Disease
Keywords: CARBIDOH
MeSH Terms: conditions — Shy-Drager Syndrome; Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Intervention Model Description: It's a monocentric, randomized, double-blind study to assess the feasibility of conducting a full-scale randomized controlled trial (RCT).
  As a cross over model study, each patient will receive the 3 ratios of the investigational drug (corresponding to the 3 arms) in a random order.
Who Masked: Participant, Investigator
Masking Description: Double blinded study: Nobody except pharmacists will know the ratios of the investigated product administrated at each visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ratio 1:10 i.e. 20 mg Carbidopa / 200 mg Levodopa (Active Comparator): This Carbidopa / Levodopa IMP ratio will be administered as a single dose, orally, at visit 1 or 2 or 3 (random order).
  Interventions: Drug: Administration of Carbidopa/levodopa
- Ratio 1:4 i.e. 50 mg Carbidopa / 200 mg Levodopa (Active Comparator): This Carbidopa / Levodopa IMP ratio will be administered as a single dose, orally, at visit 1 or 2 or 3 (random order).
  Interventions: Drug: Administration of Carbidopa/levodopa
- Ratio 1:2 i.e. 100 mg Carbidopa / 200 mg Levodopa (Experimental): This Carbidopa / Levodopa IMP ratio will be administered as a single dose, orally, at visit 1 or 2 or 3 (random order).
  Interventions: Drug: Administration of Carbidopa/levodopa

INTERVENTIONS:
Drug: Administration of Carbidopa/levodopa — Participants will perform beat-by-beat orthostatic tests (Schellong tests) before and after intake of single doses of carbidopa:levodopa combinations at 3 different ratios

SUMMARY:
This study is aimed at patients with multi-system atrophy - parkinsonian type (P-MSA) or Parkinson's disease (PD) receiving dopaminergic drugs and suffering from orthostatic hypotension (OH).

OH is a drop in blood pressure when standing, which can lead to symptoms of dizziness, lightheadedness, a black veil in front of the eyes and, when severe, can lead to fainting. HO is one of the symptoms present in AMS-P and PD.

The standard treatment for parkinsonian symptoms of slowness and stiffness is the administration of antiparkinsonian drugs containing dopamine. These dopaminergic drugs always contain 1) levodopa (which is the precursor of dopamine) and 2) an enzyme inhibitor, which may be either benserazide (in the case of Madopar® and its generics) or carbidopa (in the case of Sinemet® or Stalevo® and their generics) and whose role is to potentiate the effect of levodopa.

It has long been known that dopaminergic drugs aggravate HO. Through various mechanisms, this worsening of HO is linked as much to levodopa as to the enzyme inhibitor with which it is combined. However, investigators do not know the respective effects of these two molecules on HO.

In this study, investigators examine how the ratio of Carbidopa to levodopa affects HO in the various assays of the dopaminergic drug under study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed.
2. Patient over 18 years and under 80 years of age.
3. Patient with Multiple System Atrophy- Parkinsonian type (MSA-P) (confirmed by diagnostic criteria for clinically established and clinically probable multiple system atrophy (11); OR Patient with Parkinson Disease (PD) (12) presenting OH symptoms (getting at least one point at the 3 questions - n° 14, 15 and 16 - of the SCOPA-AUT scale that address orthostatic hypotension symptoms).
4. Patient currently receiving Dopamine-Replacement Therapy (i.e. Levodopa combined with Carbidopa or Benserazide).

Exclusion Criteria:

1. Patient unable to stand an overnight (at least 12 hours) withdrawal of their immediate-release DRT (last extended-, delayed-, or controlled-release dosage must be taken minimum 24 hours prior to the test).
2. Patient with known congestive heart failure, grades C and D, NYHA III and IV.
3. Patient with dementia (i.e. major cognitive impairment) associated to MSA-P or PD,
4. Patient with mild cognitive impairment, and unable to provide or understand informed consent, i.e. who does not have full capacity for discernment.
5. Current participation to other clinical trials.
6. Pregnant or lactating woman or willing to become pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of future large-scale double-blind randomized controlled trial (RCT) | From enrollment to the end of study at 5 weeks.
  The primary objective is to investigate the feasibility of conducting a future large-scale double-blind randomized controlled trial (RCT) assessing the effect on orthostatic hypotension (OH) of different dosages of Carbidopa (20, 50 or 100 mg), for a constant Levodopa dose (200 mg) through:
  * Recruitment rate: Mean number of patients informed per month during the recruitment period, % of patients wiling to participate to the study among the informed patients, % of patients eligible among the informed patients
  * Adherence rate:% of patients completing the study intervention period among randomized patients
  * Retention rate:% of patients showing up at the last follow-up visit among patients who have completed the study intervention period, % of drop-outs among randomized patients at last follow-up visit
  * Data completion rate of the therapeutic effect measures: % of patients with analysable OH data at week 1, 2 and 3.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Yes